CLINICAL TRIAL: NCT01924286
Title: Preventing Tuberculosis-associated Immune Reconstitution Inflammatory Syndrome in High-risk Patients: a Randomized Placebo-controlled Trial of Prednisone
Brief Title: Preventing TB-IRIS in High-risk Patients: a Randomized Placebo-controlled Trial of Prednisone
Acronym: Pred-ART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Imperial College London (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Department of Science and Technology, South Africa (Unknown)
Responsible Party: Principal Investigator, Graeme Meintjes, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIDRI_001; SP.2011.41304.074 (Other Grant/Funding Number: EDCTP); DOH-27-0813-4336 (Registry Identifier: South African National Health Research Ethics Council)
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Immune Reconstitution Inflammatory Syndrome; HIV; Tuberculosis
Keywords: HIV; Tuberculosis; Immune reconstitution inflammatory syndrome; Highly active antiretroviral therapy; Glucocorticoids; Prednisone; Preventive therapy
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; Tuberculosis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Prednisone oral tablets 40mg daily for 2 weeks followed by 20mg daily for 2 weeks
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Placebo oral tablets 40mg daily for 2 weeks followed by 20mg daily for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone
  Other Names: Trolic
  Arms: Prednisone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Tuberculosis (TB) is the most common opportunistic infection amongst HIV-infected patients starting antiretroviral therapy (ART) in developing countries and thus the most frequent form of immune reconstitution inflammatory syndrome (IRIS). Paradoxical TB-IRIS occurs in 8- 43% of patients starting ART while on TB treatment and results in morbidity, hospitalisation, consumes health care resources and TB-IRIS may be fatal. We have previously demonstrated in a clinical trial that prednisone reduces morbidity when used for treatment of paradoxical TB-IRIS. This trial is a double-blind placebo-controlled trial of prophylactic prednisone (40mg/day for 2 weeks followed by 20mg/day for 2 weeks, started on the same day as ART) in patients with TB who are identified as being at high risk for paradoxical TB-IRIS (starting ART within 30 days of initiating TB treatment and CD4 < 100/μL). The trial will enroll 240 participants, randomised 1:1 (prednisone:placebo). The primary endpoint is development of paradoxical TB-IRIS, defined using international consensus case definitions. Secondary endpoints include time to IRIS event, severity of IRIS, quality of life assessment, mortality and corticosteroids adverse events. The trial is powered to determine a reduction in TB-IRIS events.

DETAILED DESCRIPTION:
Objective: To determine whether the addition of prednisone to the first 4 weeks of antiretroviral therapy (ART) reduces the risk of paradoxical TB-IRIS in HIV-infected patients being treated for TB who are at high risk of developing TB-IRIS (CD4 <100 cells/μl and starting ART within 30 days of TB treatment).

Design: A randomized double-blind placebo-controlled trial to evaluate the incidence of paradoxical TB-IRIS over the first 12 weeks of ART in participants who receive a 4 week course of prednisone versus participants who receive a 4 week course of placebo.

Primary efficacy endpoint:

The development of paradoxical TB-IRIS within 12 weeks of starting ART (defined using the International Network for the Study of HIV-associated IRIS (INSHI) consensus case definition).

Secondary efficacy endpoints:

1. Time to IRIS event
2. Severity of IRIS events (defined by the following: need for hospitalisation for IRIS, C-reactive protein, and neurological involvement)
3. Duration of TB-IRIS event (from onset of symptoms/signs to resolution of TB-IRIS symptoms/signs)
4. Mortality attributed to TB and TB-IRIS
5. All-cause mortality
6. Composite endpoint of death, hospitalization, or hepatotoxicity (using the protocol-specified definition of Grade 3 or 4 increase in ALT or bilirubin).
7. Other (non-TB) IRIS events
8. Quality of life assessment (measured using PROQOL-HIV, EQ-5D-3L, HIV symptom index and Karnofsky score)
9. Adverse events and severe adverse events ascribed to TB treatment, ART or co-trimoxazole. This will include a pre-specified analysis of drug-induced liver injury and drug rash. This assessment will include the number of treatment interruptions for drug adverse events.
10. Discontinuation of either ART or TB treatment for > 5 days due to adverse events
11. Number of hospitalizations and total days hospitalized

Safety and tolerability endpoints:

1. Corticosteroid-associated adverse events, classified by severity and relation to study drug. These will include hypertension, hyperglycaemia, hypomania/mania, depression, acne, epigastric pain, upper gastro-intestinal bleeding, Cushingoid features, new oedema and avascular bone necrosis.
2. Laboratory safety data: glucose, full blood count and electrolytes
3. Other infections (AIDS-related, bacterial, fungal and viral) and malignancies (Kaposi's sarcoma)
4. All grade 1, 2, 3 and 4 adverse events (clinical and laboratory using the ACTG grading system)

Sample size: 240 participants will be enrolled over 13 months. Each participant will be followed for 12 weeks.

Population: HIV-infected, ART-naïve adult (≥ 18 years) patients diagnosed with active tuberculosis who have a CD4 < 100 cells/μL and who start ART within 30 days of starting TB treatment. Other inclusion criteria include: diagnosis of TB (smear, culture, Xpert MTB/RIF test, histology or strong clinical and radiological evidence of TB with symptomatic response to TB treatment), eligible for and consent to starting ART and written informed consent for trial. Exclusion criteria include: Kaposi's sarcoma, pregnancy, TB meningitis or tuberculoma at TB diagnosis (because these patients receive corticosteroids), known rifampicin-resistant TB, being on corticosteroids for another indication within the past 7 days, on other immunosuppressive medication within the past 7 days and uncontrolled diabetes mellitus.

TB treatment and ART: TB treatment will be prescribed and monitored by the clinical staff in the local HIV-TB clinic. TB treatment will be given according to South African Department of Health guidelines. This involves rifampicin (R), isoniazid (H), ethambutol (E) and pyrazinamide (Z) for 2 months followed by RH for 4 months. ART will be prescribed by the clinical staff at the HIV-TB clinic according to South African Department of Health guidelines. Standard first line ART in TB patients is tenofovir, emtricitabine (or lamivudine) and efavirenz. Co-trimoxazole prophylaxis will be prescribed to all patients unless a contra-indication exists.

Intervention: Oral prednisone 40mg daily for 14 doses started on the first day that ART is taken, followed by 20mg daily for 14 doses (or identical placebo). A total of 28 days of study medication will thus be prescribed.

Follow-up: Patients will be screened once established on TB treatment, but before starting ART. If the patient is eligible, written informed consent will be taken. There will be six planned study visits that will be in relation to the start of ART: week 0 (the day ART is initiated), week 1, week 2, week 4, week 8 and week 12. Patients will be seen at unscheduled visits if clinical deterioration occurs. If paradoxical TB-IRIS is diagnosed this will be treated with open label prednisone at clinician discretion if symptoms are moderate or severe. If patients experience clinical complications (eg. TB-IRIS) follow-up will be prolonged beyond week 12 in order to stabilize their condition before referral back to the general TB-HIV clinical service for ongoing management.

Data monitoring: The trial will be monitored by an independent Data and Safety Monitoring Board (DSMB) comprising 3 independent researchers and an independent statistician. After an initial meeting for agreeing on their Charter, the DSMB will meet twice (after 80 and 160 participants have completed follow-up) to review data quality and data with respect to safety and trial endpoints. If there is evidence of harm related to study medication or trial conduct the DSMB may advise the sponsor that trial enrollment should be stopped.

Clinical trial site: Khayelitsha Site B HIV-TB clinic (Ubuntu clinic)

Co-investigators:

Lut Lynen (Institute of Tropical Medicine, Antwerp, Belgium) Gary Maartens (University of Cape Town) Robert J. Wilkinson (Imperial College London and University of Cape Town) Robert Colebunders (Institute of Tropical Medicine, Antwerp, Belgium)

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected HIV infection will be confirmed by two different rapid tests (as per South African national Department of Health guidelines) and an HIV viral load test.
2. CD4 count < 100/μL One CD4 count taken within 3 months prior to enrolment less than 100/μL will qualify, even if other CD4 counts are greater than 100/μL
3. ART-naïve Patients who report having been treated with triple drug or dual drug ART previously will be excluded. Single dose nevirapine or short term AZT monotherapy for PMTCT is not an exclusion.
4. Confirmed diagnosis of TB (smear, culture, Xpert MTB/RIF test or compatible histology) or strong clinical and radiological evidence of TB with symptomatic response to TB treatment
5. On TB treatment for less than 30 days prior to study entry.
6. Eligible for ART and patient consents to starting ART within 30 days of starting TB treatment.
7. Written informed consent for trial

Exclusion Criteria:

1. Kaposi's sarcoma (KS) A thorough examination for KS lesions will be performed and any suspicious lesion will be biopsied. Any history of treatment for KS will also be an exclusion.
2. Pregnant All female participants of child-bearing potential will have a pregnancy test performed prior to enrollment and will be counseled to use to two reliable methods of contraception for the duration of the trial.
3. <18 years old
4. TB meningitis or tuberculoma at TB diagnosis
5. Clinical syndrome of pericardial TB at TB diagnosis (a pericardial effusion noted on ultrasound scan alone is not an exclusion criterion)
6. Rifampicin-resistant TB diagnosed by Xpert MTB/RIF test or a drug susceptibility test performed on a culture isolate.
7. On corticosteroids for another indication or on any other immunosuppressive medication within the past 7 days.
8. Uncontrolled diabetes mellitus
9. The following abnormal laboratory values:

   Alanine aminotransferase > 200 IU/l Absolute neutrophil count < 500/mm3
10. Not on standard intensive phase TB treatment (Rifampicin, isoniazid, pyrazinamide and ethambutol)
11. Poor clinical response to TB treatment prior to ART as judged by the clinical investigators.
12. Hepatitis B surface antigen positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Development of paradoxical TB-IRIS | 12 weeks
  The development of paradoxical TB-IRIS within 12 weeks of starting ART (defined using the International Network for the Study of HIV-associated IRIS (INSHI) consensus case definition)

SECONDARY OUTCOMES:
Time to IRIS event | 12 weeks
Severity of IRIS events | 12 weeks
  Defined by the following: need for hospitalisation for IRIS, C-reactive protein, and neurological involvement
Duration of TB-IRIS event | Average 8-12 weeks from onset
  From onset of symptoms/signs to resolution of TB-IRIS symptoms/signs. Participants will be followed until resolution of TB-IRIS symptoms/signs which is an average 8-12 weeks from onset.
Mortality attributed to TB and TB-IRIS | 12 weeks
All-cause mortality | 12 weeks
Composite endpoint of death, hospitalization, or hepatotoxicity (using the protocol-specified definition of Grade 3 or 4 increase in ALT or bilirubin) | 12 weeks
Other (non-TB) IRIS events | 12 weeks
  Number of other IRIS events (other than TB-IRIS) occurring in participants
Adverse events and severe adverse events ascribed to TB treatment, ART or co-trimoxazole | 12 weeks
  This will include a pre-specified analysis of drug-induced liver injury and drug rash. This assessment will include the number of treatment interruptions for drug adverse events.
Discontinuation of either ART or TB treatment for > 5 days due to adverse events | 12 weeks
Number of hospitalizations | 12 weeks
Corticosteroid-associated adverse events, classified by severity and relation to study drug | 12 weeks
  These will include hypertension, hyperglycaemia, hypomania/mania, depression, acne, epigastric pain, upper gastro-intestinal bleeding, Cushingoid features, new oedema and avascular bone necrosis
Laboratory safety data: Glucose | 12 weeks
Other infections (AIDS-related, bacterial, fungal and viral) and malignancies (Kaposi's sarcoma) | 12 weeks
All grade 1, 2, 3 and 4 adverse events (clinical and laboratory using the ACTG grading system) | 12 weeks
Total number of days hospitalised | 12 weeks
Laboratory safety data: Haemoglobin | 12 weeks
Laboratory safety data: White cell count | 12 weeks
Laboratory safety data: Serum sodium | 12 weeks
Laboratory safety data: Serum potassium | 12 weeks

OTHER OUTCOMES:
Quality of life assessment | 12 weeks
  Quality of life assessment (measured using PROQOL-HIV)
Quality of life assessment | 12 weeks
  Measured using EQ-5D-3L
Quality of life assessment | 12 weeks
  Measured using HIV symptom index
Quality of life assessment | 12 weeks
  Measured using Karnofsky score

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Meintjes, MD MPH PhD, Principal Investigator — University of Cape Town
Locations (1):
- Site B Khayelitsha HIV/TB clinic, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Meintjes G, Stek C, Blumenthal L, Thienemann F, Schutz C, Buyze J, Ravinetto R, van Loen H, Nair A, Jackson A, Colebunders R, Maartens G, Wilkinson RJ, Lynen L; PredART Trial Team. Prednisone for the Prevention of Paradoxical Tuberculosis-Associated IRIS. N Engl J Med. 2018 Nov 15;379(20):1915-1925. doi: 10.1056/NEJMoa1800762. PMID 30428290